CLINICAL TRIAL: NCT00813189
Title: Effects of Growth Hormone on Corticoid Myopathy in Children With Chronic Disease: Effects on Muscle Mass and Strength
Brief Title: Efficacy Study of Recombinant Growth Hormone on Muscle Function in Children Long-term Treated With Glucocorticoid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association REMEDE (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dominique SIMON, dominique Simon MD, Association REMEDE
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004/64
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Disease; Glucocorticoid Therapy, Response to; Growth Retardation
Keywords: glucocorticoid therapy; muscle function; growth hormone treatment
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 : early start (GH treatment) group (Experimental): in the early start group, patients were treated with growth hormone for one year immediately after randomisation
  Interventions: Device: GH treatment
- 2 :delayed start (GH treatment) group (No Intervention): in the delayed start group patients took GH treatment for 1 year , 6 months after randomisation

INTERVENTIONS:
Device: GH treatment — GH treatment will be administered at a weekly dose of 0.46 mg/kg/ week, divided into seven daily subcutaneous injections. Subcutaneous injections should be given slowly, in the thigh. In order to prevent lipoatrophy, the injection site should be varied. The injection should be given at bedtime.
  Arms: 1 : early start (GH treatment) group

SUMMARY:
Children suffering from chronic disease and receiving long-term glucocorticoid therapy suffer over years from severe growth retardation and profoundly altered body composition. They consist in a marked increase in fat mass and a decrease in lean body mass. Published studies have shown that Growth Hormone (GH) treatment in children with Juvenile Idiopathic Arthritis can improve body composition by increasing lean mass and by preventing increase in fat mass. The aim of the present protocol is to evaluate whether the increase in lean body mass observed during GH treatment is associated with changes in muscle strength and mass.

In order to be able to evaluate the effect of GH on the muscle a comparative group is needed. Therefore it will be proposed to delay in a group of patients the start of Growth Hormone(GH) treatment by 6 months. As most publications have shown a maximum effect of GH within the first year of treatment, six months should be enough to evaluate short-term effect of GH on the muscle. Therefore, this study will be a randomized trial: immediate start of Growth Hormone (GH) treatment versus start of Growth Hormone treatment 6 months later. After 6 months all children will be treated with GH. Therefore, the follow-up will be one year after baseline.

DETAILED DESCRIPTION:
The aim of the present protocol is to evaluate the effects of GH treatment in long-term steroid treated children, on muscle mass, and muscle strength. It will be an open, randomized, controlled, 2-parallel group study. The follow-up in this study will be one year. The objective of this study will be to evaluate short-term effects of GH treatment on muscle mass, muscle strength and body composition in children suffering from various diseases requiring steroid therapy. Expected pathologies are juvenile idiopathic arthritis, nephrotic syndrome, uveitis, systemic diseases and organ transplantation. Changes in muscle mass will be assessed by measuring the muscle and sub-cutaneous fat on the cross sectional area of the thigh by MRI. MRI offer the advantage of non-invasive technique, allowing serial and accurate measurements.Muscle strength will be performed by serial muscular testing of different muscular groups. Body composition will be assessed by DEXA. DEXA allows rapid, accurate and highly reproductible determination not only of bone mass but also of lean and fat mass of the whole body, with very low radiation exposure.It appears to be the most sensitive method for assessment of muscle wasting as well as of fat repartition that contribute to Cushing's appearance in steroid treated patients.

The present study will be performed in children with growth retardation related to long-term glucocorticoid treatment These patients had never been treated with GH. In order to be able to evaluate the effect of GH on the muscle a comparative group is needed. Therefore it will be proposed in the study to delay in a group of patient the start of GH treatment by 6 months. Six months should be enough to evaluate short-term effect of GH on the muscle and most publication have shown a maximum effect of GH within the first year of treatment. Therefore, this study will be a randomized trial: immediate start of GH treatment versus start of GH treatment 6 months later. After 6 months all children will be treated with GH. The dose administered in the present trial will be a GH dose already tested in glucocorticoid treated children (0.46 mg/kg/week)

ELIGIBILITY:
Inclusion Criteria:

* Measured Height below -2 SD
* Bone age below 13 years for a boy and below 11 years for a girl
* Glucocorticosteroid treatment for 12 months at least
* Glucocorticosteroid dose above or equal to 0.2 mg/kg/day of prednisone or equivalent dose over the last 12 months
* Glucocorticosteroid treatment is anticipated to be sustained for 1 more year at least
* The child benefits of the French social security cover
* Child who has never been treated by GH.
* Evidence of a personally signed and dated informed consent document indicating that the patient's parents/guardians and from the patient himself/herself if he/she is able to receive and understand the information have been informed of all pertinent aspects of the study.
* No glucose intolerance or diabetes mellitus on an Oral Glucose Tolerance Test dated less than 3 months

Exclusion Criteria:

* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-04; Primary Completion 2010-06 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The main criteria of efficacy will be - the mean strength changes assessed as a composite score (mean of the relative changes of the ten muscle functions tested): ∆ strength as % of baseline values :6 months-baseline. | 6 months

SECONDARY OUTCOMES:
Strength changes assessed as a composite score (mean of the relative changes of the ten muscle functions tested) as % of baseline values : 12 months-baseline and 12 months- 6 months, 18 months- 6 months for group B patients | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique SIMON, PHD, Principal Investigator — Hopital Robert -Debré, Assistance Publique, Hopitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France